CLINICAL TRIAL: NCT05842096
Title: The Influence of Subclinical Hypothyroidism on Chronic Inflammation Activity in Women With Different PCOS Phenotypes
Brief Title: Subclinical Hypothyroidism and Chronic Inflammation in PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, Ph.D., Principal Investigator, Jagiellonian University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1072.6120.292.2022
Record Dates: First submitted 2023-03-26; First posted 2023-05-03 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries; Subclinical hypothyroïdism; Hypothalamic-Pituitary-Gonadal Axis Dysfunction
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: prospective tertiary single-centre cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polycystic ovary syndrome (PCOS) (Active Comparator): Women meeting the Rotterdam-ESHRE-ASRM criteria for a diagnosis of PCOS
  Interventions: Diagnostic Test: Measurement and comparison of leucocytosis and concentrations of CRP, procalcitonin, fibrinogen, ferritin, IL-1, IL-6, IL-10, TNF-alpha in both study arms; Diagnostic Test: Evaluation of the impact of subclinical hypothyroidism, with present/ absent antithyroid antibodies, on the balance between anti- and pro-inflammatory factors in women in both study arms; Diagnostic Test: Assessment of the impact of imbalance between anti- and pro-inflammatory factors in women with different PCOS and HPOD phenotypes on ovarian reserve indices
- Hypothalamic-Pituitary-Ovarian Axis Dysfunction (HPOD) (Active Comparator): Women meeting the WHO criteria for a diagnosis of HPOD
  Interventions: Diagnostic Test: Measurement and comparison of leucocytosis and concentrations of CRP, procalcitonin, fibrinogen, ferritin, IL-1, IL-6, IL-10, TNF-alpha in both study arms; Diagnostic Test: Evaluation of the impact of subclinical hypothyroidism, with present/ absent antithyroid antibodies, on the balance between anti- and pro-inflammatory factors in women in both study arms; Diagnostic Test: Assessment of the impact of imbalance between anti- and pro-inflammatory factors in women with different PCOS and HPOD phenotypes on ovarian reserve indices

INTERVENTIONS:
Diagnostic Test: Measurement and comparison of leucocytosis and concentrations of CRP, procalcitonin, fibrinogen, ferritin, IL-1, IL-6, IL-10, TNF-alpha in both study arms — A venous blood sample of approximately 10 ml will be collected in the morning after 8 hours of fasting to determine and compare the above parameters of peripheral blood in both arms of the study
Diagnostic Test: Evaluation of the impact of subclinical hypothyroidism, with present/ absent antithyroid antibodies, on the balance between anti- and pro-inflammatory factors in women in both study arms — A venous blood sample of approximately 10 ml will be collected in the morning after 8 hours of fasting to determine and compare blood levels of leukocytosis, CRP, procalcitonin, fibrinogen, ferritin, IL-1, IL-6, IL-10, TNF-alpha depending on the blood concentrations of TSH, a-TPO and a-TG in women in both study arms
Diagnostic Test: Assessment of the impact of imbalance between anti- and pro-inflammatory factors in women with different PCOS and HPOD phenotypes on ovarian reserve indices — A venous blood sample of approximately 10 ml will be collected in the morning after 8 hours of fasting to determine and compare blood levels of leukocytosis, CRP, procalcitonin, fibrinogen, ferritin, IL-1, IL-6, IL-10, TNF-alpha and AMH, FSH in women in both study arms

SUMMARY:
Chronic inflammation in polycystic ovary syndrome (PCOS) may be the result of dysregulation of cytokine production (due to insulin resistance, excess visceral fat and hyperandrogenemia), i.e., overproduction of pro-inflammatory factors (e.g. TNF, IL-1, IL-6) in relation to anti-inflammatory ones (IL-10). This condition may be an important link between obesity and insulin resistance, which is crucial in the etiopathogenesis of the syndrome. However, it is not known whether it results from the tendency to accumulate adipose tissue or is a feature of the syndrome itself. Concomitant endocrinopathies, i.e. obesity, dyslipidemia, insulin resistance, diabetes and thyroid diseases, may additionally influence the activity of chronic inflammation. There is no data indicating the relationship between chronic inflammation and PCOS phenotypes, the severity of metabolic disorders, ovarian reserve and the influence of thyroid function on its activity in PCOS.

DETAILED DESCRIPTION:
The aim of the study is:

i) to assess and compare serum concentrations of selected inflammatory markers (leucocytosis, CRP, procalcitonin, fibrinogen, ferritin, IL-1, IL-6, IL-10, TNF-alpha) in women with different phenotypes PCOS and hypothalamic-pituitary-ovarian axis dysfunction (HPOD) (control), ii) to evaluate the impact of subclinical hypothyroidism (defined as TSH>2.5 uIU/ml, fT3 3,1-6,80 pmol/l, fT4 12,0-22,0 pmol/l), with the presence and absence of circulating antithyroid antibodies (a-TPO and a-TG), on the balance between anti- and pro-inflammatory factors in women with different PCOS and HPOD phenotypes, iii) to assess the impact of imbalance between anti- and pro-inflammatory factors in women with different PCOS and HPOD phenotypes on ovarian reserve indices, expressed as FSH and AMH concentrations.

The study population will be characterized in terms of demographic (age, BMI), gynecological (age of first and last menstrual period, cycle length, history of reproductive organ surgeries, ultrasound measurements of endometrial width, ovarian volume) and obstetrics (pregnancies, childbirth, miscarriages) data. PCOS syndrome (and its phenotypes) will be recognized by the Rotterdam criteria. HPOD will be diagnosed according to WHO criteria. During hospitalization, blood samples will be collected for scheduled analyzes (30 ml of blood in total).

ELIGIBILITY:
Inclusion Criteria:

* age 18-45 years,
* cycle length <21 days or > 35 days,
* unsuccessful attempts to conceive for at least 12 months of regular intercourse with sonographically confirmed anovulation with excluded male, tubal and uterine infertility factors.

Exclusion Criteria:

* absence of at least one ovary,
* previously diagnosed thyroid disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Values of inflammation parameters - leukocytosis in peripheral blood in both study arms | up to 6 months
  Measurement and comparison of leukocyte count (n/µL) in peripheral blood in both study arms
Values of inflammation parameters - CRP in peripheral blood in both study arms | up to 6 months
  Measurement and comparison of concentrations of CRP (mg/l) in peripheral blood in both study arms
Values of inflammation parameters - procalcitonine in peripheral blood in both study arms | up to 6 months
  Measurement and comparison of concentrations of procalcitonin (μg/l) in peripheral blood in both study arms
Values of inflammation parameters - fibrinogen in peripheral blood in both study arms | up to 6 months
  Measurement and comparison of concentrations of procalcitonin fibrinogen (g/l) in peripheral blood in both study arms
Values of inflammation parameters - ferritin in peripheral blood in both study arms | up to 6 months
  Measurement and comparison of concentrations of procalcitonin ferritin (μg/l) in peripheral blood in both study arms
Values of inflammation parameters - IL-1 in peripheral blood in both study arms | up to 6 months
  Measurement and comparison of concentrations of procalcitonin IL-1 (pg/ml) in peripheral blood in both study arms
Values of inflammation parameters - IL-6 in peripheral blood in both study arms | up to 6 months
  Measurement and comparison of concentrations of procalcitonin IL-6 (pg/ml) in peripheral blood in both study arms
Values of inflammation parameters - IL-10 in peripheral blood in both study arms | up to 6 months
  Measurement and comparison of concentrations of procalcitonin IL-10 (pg/ml) in peripheral blood in both study arms
Values of inflammation parameters - TNF-alpha in peripheral blood in both study arms | up to 6 months
  Measurement and comparison of concentrations of procalcitonin TNF-alpha (pg/ml) in peripheral blood in both study arms

SECONDARY OUTCOMES:
Correlation between the concentration of TSH (mIU/l) and the parameters of inflammation - leukocytosis in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of TSH (mIU/l) and inflammatory parameters: leukocyte count (n/µL)
Correlation between the concentration of TSH (mIU/l) and the parameters of inflammation - CRP in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of TSH (mIU/l) and inflammatory parameters: CRP (mg/l)
Correlation between the concentration of TSH (mIU/l) and the parameters of inflammation - procalcitonin in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of TSH (mIU/l) and inflammatory parameters: procalcitonin (μg/l)
Correlation between the concentration of TSH (mIU/l) and inflammatory parameters: fibrinogen (μg/l) | up to 6 months
  Evaluation of the correlation between the concentration of TSH (mIU/l) and inflammatory parameters: fibrinogen (g/l)
Correlation between the concentration of TSH (mIU/l) and inflammatory parameters: ferritin (μg/l) | up to 6 months
  Evaluation of the correlation between the concentration of TSH (mIU/l) and inflammatory parameters: ferritin (μg/l)
Correlation between the concentration of TSH (mIU/l) and inflammatory parameters: il-1 | up to 6 months
  Evaluation of the correlation between the concentration of TSH (mIU/l) and inflammatory parameters: iL-1 (pg/ml)
Correlation between the concentration of TSH (mIU/l) and inflammatory parameters: il-6 | up to 6 months
  Evaluation of the correlation between the concentration of TSH (mIU/l) and inflammatory parameters: iL-6 (pg/ml)
Correlation between the concentration of TSH (mIU/l) and inflammatory parameters: il-10 | up to 6 months
  Evaluation of the correlation between the concentration of TSH (mIU/l) and inflammatory parameters: iL-10 (pg/ml)
Correlation between the concentration of TSH (mIU/l) and inflammatory parameters: TNF-alpha | up to 6 months
  Evaluation of the correlation between the concentration of TSH (mIU/l) and inflammatory parameters: TNF-alpha (pg/ml)
Correlation between the concentration of a-TPO (IU/ml) and the parameters of inflammation - leukocytosis in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: leukocyte count (n/µL)
Correlation between the concentration of a-TPO (IU/ml) and the parameters of inflammation - CRP in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: CRP (mg/l)
Correlation between the concentration of a-TPO (IU/ml) and the parameters of inflammation - procalcitonin in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: procalcitonin (μg/l)
Correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: fibrinogen (μg/l) | up to 6 months
  Evaluation of the correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: fibrinogen (μg/l)
Correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: ferritin (μg/l) | up to 6 months
  Evaluation of the correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: ferritin (μg/l)
Correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: il-1 (pg/ml) | up to 6 months
  Evaluation of the correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: il-1 (pg/ml)
Correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: il-6 (pg/ml) | up to 6 months
  Evaluation of the correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: il-6 (pg/ml)
Correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: il-10 (pg/ml) | up to 6 months
  Evaluation of the correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: il-10 (pg/ml)
Correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: TNF-alpha (pg/ml) | up to 6 months
  Evaluation of the correlation between the concentration of a-TPO (IU/ml) and inflammatory parameters: TNF -alpha (pg/ml)
Correlation between the concentration of a-TG (IU/ml) and the parameters of inflammation - CRP in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: CRP (mg/l)
Correlation between the concentration of a-TG (IU/ml) and the parameters of inflammation - leukocytosis in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: leukocyte count (n/µL)
Correlation between the concentration of a-TG (IU/ml) and the parameters of inflammation - procalcitonin in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: procalcitonin (μg/l)
Correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: fibrinogen (μg/l) | up to 6 months
  Evaluation of the correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: fibrinogen (μg/l)
Correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: il-1 (pg/ml) | up to 6 months
  Evaluation of the correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: il-1 (pg/ml)
Correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: il-6 (pg/ml) | up to 6 months
  Evaluation of the correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: il-6 (pg/ml)
Correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: il-10 (pg/ml) | up to 6 months
  Evaluation of the correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: il-10 (pg/ml)
Correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: TNF-alpha (pg/ml) | up to 6 months
  Evaluation of the correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: TNF-alpha (pg/ml)
Correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: ferritin (μg/l) | up to 6 months
  Evaluation of the correlation between the concentration of a-TG (IU/ml) and inflammatory parameters: ferritin (μg/l)
Correlation between the concentration of AMH (pmol/l) and the parameters of inflammation - leukocytosis in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of AMH (pmol/l) and inflammatory parameters: leukocyte count (n/µL)
Correlation between the concentration of AMH (pmol/l) and the parameters of inflammation - CRP in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of AMH (pmol/l) and inflammatory parameters: CRP (mg/l)
Correlation between the concentration of AMH (pmol/l) and the parameters of inflammation - procalcitonin in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of AMH (pmol/l) and inflammatory parameters: procalcitonin (μg/l)
Correlation between the concentration of AMH (pmol/l) and the parameters of inflammation - fibrinogen in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of AMH (pmol/l) and inflammatory parameters: fibrinogen (μg/l)
Correlation between the concentration of AMH (pmol/l) and the parameters of inflammation - ferritin in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of AMH (pmol/l) and inflammatory parameters: ferritin (μg/l)
Correlation between the concentration of AMH (pmol/l) and the parameters of inflammation - il-1 in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of AMH (pmol/l) and inflammatory parameters: il-1 (pg/ml)
Correlation between the concentration of AMH (pmol/l) and the parameters of inflammation - il-6 in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of AMH (pmol/l) and inflammatory parameters: il-6 (pg/ml)
Correlation between the concentration of AMH (pmol/l) and the parameters of inflammation - il-10 in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of AMH (pmol/l) and inflammatory parameters: il-10 (pg/ml)
Correlation between the concentration of AMH (pmol/l) and the parameters of inflammation - TNF-alpha in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of AMH (pmol/l) and inflammatory parameters: TNF-alpha (pg/ml)
Correlation between the concentration of FSH (IU/l) and the parameters of inflammation - leukocytosis in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of FSH (IU/l) and inflammatory parameters: leukocyte count (n/µL)
Correlation between the concentration of FSH (IU/l) and the parameters of inflammation - CRP in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of FSH (IU/l) and inflammatory parameters: CRP (mg/l)
Correlation between the concentration of FSH (IU/l) and the parameters of inflammation - procalcitonin in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of FSH (IU/l) and inflammatory parameters: procalcitonin (μg/l)
Correlation between the concentration of FSH (IU/l) and the parameters of inflammation - fibrinogen in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of FSH (IU/l) and inflammatory parameters: fibrinogen (μg/l)
Correlation between the concentration of FSH (IU/l) and the parameters of inflammation - ferritin in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of FSH (IU/l) and inflammatory parameters: ferritin (μg/l)
Correlation between the concentration of FSH (IU/l) and the parameters of inflammation - il-1 in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of FSH (IU/l) and inflammatory parameters: il-1 (pg/ml)
Correlation between the concentration of FSH (IU/l) and the parameters of inflammation - il-6 in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of FSH (IU/l) and inflammatory parameters: il-6 (pg/ml)
Correlation between the concentration of FSH (IU/l) and the parameters of inflammation - il-10 in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of FSH (IU/l) and inflammatory parameters: il-10 (pg/ml)
Correlation between the concentration of FSH (IU/l) and the parameters of inflammation - TNF-alpha in both arms of the study | up to 6 months
  Evaluation of the correlation between the concentration of FSH (IU/l) and inflammatory parameters:TNF-alpha (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jach, Prof., Ph.D., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Department of Gynecology and Obstetrics, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No